CLINICAL TRIAL: NCT04844034
Title: The Effects of a High Eicosapentaenoic Acid Multinutrient Supplement on Measures of Stress, Anxiety and Depression in Young Adults: a Randomised, Double-blind, Placebo-controlled Trial.
Brief Title: Effects of a High EPA Multinutrient Supplement on Negative Affect in Young Adults.
Acronym: NutriMOOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roehampton (Other)
Responsible Party: Principal Investigator, Dr Simon Dyall, Dr, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SD001
Record Dates: First submitted 2021-03-16; First posted 2021-04-14 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Anxiety; Depression
Keywords: Anxiety; Depression; Anxiolytic; Antidepressant; Omega-3 PUFAs; Eicosapentaenoic Acid; Docosahexaenoic Acid; Long-chain Polyunsaturated Fatty Acids; Dietary Supplement; Stress; Functional magnetic resonance imaging; Magnetic resonance spectroscopy
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator): High-EPA multinutrient supplement.
  Interventions: Dietary Supplement: High-EPA multinutrient supplement.
- Placebo (Placebo Comparator): Inert oil mix.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: High-EPA multinutrient supplement. — Three capsules with the largest meal of the day providing:
  * 1,125 mg EPA
  * 441 mg DHA
  * 330 mg Magnesium
  * 7.5 mg a-tocopherol
  Other Names: Libretto
  Arms: Active treatment
Other: Placebo — Three capsules with the largest meal of the day providing:
  * 3,060 mg sunflower seed oil
  * 60 mg lecithin
  * 300 mg glyceryl monostearate
  * 465 mg EPA/DHA (18%/12% respectively for blinding)
  Arms: Placebo

SUMMARY:
This is a 12-week-long, randomised, double-blind, placebo-controlled trial exploring the efficacy of a high-EPA multinutrient supplement in the management of sub-clinical anxiety and depression. The investigators focus on young and healthy, adult university students, who may otherwise not be eligible for pharmacological or cognitive behavioural therapy interventions.

DETAILED DESCRIPTION:
First-line treatment for anxiety disorders comprises Cognitive Behavioural Therapy, which is ineffective in a considerable minority of individuals, and pharmacological treatments, which often confer significant side effects. On the other hand, fish-oil-based supplements have been shown to be safer, efficacious alternatives, especially for individuals not eligible for behavioural or pharmacological therapies. Evidence from randomised controlled trials (RCTs) suggests that the long-chain omega-3 polyunsaturated fatty acids (LCn-3 PUFAs) eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) may exert beneficial anxiolytic effects. It is also suggested that dietary components such as vitamins and minerals e.g. a-tocopherol (vitamin E) and Magnesium (Mg), may also play a role in mood. It is furthermore theorised that minor allelic carriage of desaturase and apolipoprotein E (APOE) polymorphisms may also influence the putative anxiolytic potential of dietary components. However, despite the abundance of findings in RCTs and animal studies, the putative synergism, additive effects and precise mechanism of action of these macro- and micronutrients on anxiety in humans are largely unknown. Furthermore, the evidence suggests that in depressive states, glutamate homeostasis is dysregulated in frontal brain regions, and in bipolar patients, glutamate concentration is increased in the anterior cingulate cortex. Supplementation with EPA-rich regimes for 12 weeks confers beneficial changes in glutamate concentrations and improvement in functional connectivity between brain regions associated with mood and improvement in global symptoms.

The investigators have designed a randomised, double-blind, placebo-controlled trial to explore the above. Students from the University of Roehampton, aged 18-29 years (Emerging Adulthood), are randomised on a 1:1 allocation ratio, in two groups, for 12 weeks:

1. Active treatment group to be supplemented with a high-EPA multinutrient supplement providing a daily dose of 1,125 mg EPA, 441 mg DHA, 330 mg magnesium and 7.5 mg α-tocopherol.
2. Placebo group to be supplemented with an inert oil mix providing a daily dose of 3,060 mg sunflower seed oil, 60 mg lecithin, 300 mg glyceryl monostearate and 465 mg fish-oil (18%/12% EPA/DHA respectively) for blinding.

Brain hemodynamic and neurochemical changes in response to supplementation with the EPA-rich regime are explored in a subgroup of volunteers by magnetic resonance imaging (MRI). Analyses take place at the Combined Universities Brain Imaging Centre (CUBIC), Royal Holloway, University of London and comprise:

1. Proton Magnetic resonance spectroscopy (MRS), to assess changes in glutamate concentrations in the right and left ventrolateral prefrontal cortex and the anterior cingulate cortex.
2. Functional MRI (fMRI) to assess changes in seed-to-voxel functional connectivity using bilateral orbitofrontal cortex (OFC) and amygdala (AMY) seeds; regions in the brain implicated in the control of emotion and mood.

The choice of the population was made on the basis of its high-risk nature; university students in Emerging Adulthood (18-29 years of age) experience persistent levels of high-academic stress, social disconnection and sleep disruption which increase anxiety levels and exacerbate psychological distress and disengagement from study. University students are thus a high-risk, vulnerable group characterised by higher and increasing rates of anxiety disorders compared to the general population. Furthermore, this population is largely neglected by the therapeutic literature.

The study hypothesis is that:

* Generally healthy, non-clinically anxious university students in Emerging Adulthood experiencing sub-clinical levels of anxiety, will benefit from supplementation with a high-EPA multinutrient supplement, in that the latter will exert beneficial anxiolytic effects.
* Mg and vitamin E will exert additive anxiolytic effects.
* Interindividual variations in fatty acid desaturases (FADS) and APOE genotypes will influence the putative anxiolytic potential of the high-EPA multinutrient supplement under investigation.
* Prefrontal and anterior cingulate cortex glutamate concentrations, and functional connectivity between OFC and AMY, will improve in response to supplementation.

The investigators will perform mixed-model analysis of covariance for the study primary and secondary endpoints, on an intention-to-treat (ITT) and per-protocol (PP) basis. The investigation which will take place at the Department of Life Sciences of the University of Roehampton and the Combined Universities Brain Imaging Centre (CUBIC), Royal Holloway, University of London, harmonised with local and national guidelines and risk assessments, the code of Good Clinical Practice and the Declaration of Helsinki. The study findings will be reported in accordance with the CONSORT statement.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-29 years
* GAD-7 Score ≥ 5
* PHQ-8 Score ≥ 4
* English language fluency.
* Overall good health.

Exclusion Criteria:

* Self reported BMI ≥ 30 kg/m^2.
* Current tobacco smoker.
* Diagnosis of anxiety, depression/major depressive disorder episode, psychosis, schizophrenia, bipolar disorder, eating disorders, haemophilia, or life-threatening disease during the preceding six months from the beginning of the trial.
* Use of antidepressant drugs during the preceding six months from the beginning of the trial.
* Participation to psychological and/or behavioural interventions during the preceding six months from the beginning of the trial.
* Inability to ingest pills.
* Pregnancy.
* Breastfeeding.
* Known allergy or intolerance to LCn-3 PUFAs, seafood and any of the constituents of the supplement under investigation.
* High intake (more than twice per week) of oily fish (e.g. herring, pilchards, salmon, swordfish, sardines, sprats, trout or mackerel).
* Use of fish oil supplements during the preceding six months from the beginning of the trial.
* Inability to participate in the study for 12 consecutive weeks.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Anxiety on the 21-point Generalised Anxiety Disorder Assessment (GAD-7) at Week 12. | Baseline and Week 12.
  GAD-7 is a 7-item, validated, self-reported instrument used to screen for generalised anxiety disorder and to assess its severity over the past two weeks. Possible scores range from 0 (none) to 21 (severe).

SECONDARY OUTCOMES:
Change from Baseline in Depression on the 24-point Patient Health Questionnaire (PHQ-8) at Week 12. | Baseline and Week 12.
  PHQ-8 is an 8-item, validated, self-reported instrument used as a diagnostic and severity measure for depressive disorders. Possible scores range from 0 (none) to 24 (severe).
Change from Baseline in Depression, Anxiety and Stress on the 21-item Depression, Anxiety and Stress Scale (DASS-21) at week 12. | Baseline and Week 12.
  DASS-21 is a validated tool comprising three self-report scales designed to measure the emotional states of depression, anxiety and stress.
Change from Baseline in the Proportion of Trials Selected as Happy Compared to the Alternative Emotion, Adjusted to a Scale of 0 to 15 on the Emotional Bias Task (EBT) at Week 12. | Baseline and Week 12.
  EBT is a 4-minute-long, computer-based test that detects perceptual bias in facial emotion perception. The key outcome measure for the EBT is the bias point; the proportion of trials selected as happy compared to the alternative emotion, adjusted to a scale of 0 to 15. This is used to determine the extent and direction of the participant's bias. Additionally, latency measures and measures of how many times each emotion was selected are also available.
Change from Baseline in Measures of Sustained Attention on the Rapid Visual Information Processing (RVP) at Week 12. | Baseline and Week 12.
  RVP is a 7-minute-long, computer-based test measuring sustained attention. Outcome measures cover latency (speed of response), probability of false alarms and sensitivity.
Change from Baseline in Measures of Retention and Manipulation of Visuospatial Information on Spatial Working Memory (SWM) at Week 12. | Baseline and Week 12.
  SWM is a 4-minute-long, computer-based test that measures strategy and working memory errors as a measure of retention and manipulation of visuospatial information. Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes which have already been found to contain a token) and strategy.
Change from Baseline in Measures of Response Inhibition on Stop Signal Task (SST) at Week 12. | Baseline and Week 12.
  SST is an up-to 14-minute-long, computer based test that measures response inhibition (impulse control). Outcome measures cover direction errors, proportion of successful stops, reaction time on Go trials, and stop signal reaction time (SSRT).

OTHER OUTCOMES:
Change from Baseline in Dietary Protein on 24-hour Dietary Intake Recall at Week 12. | Baseline and Week 12.
  Intake24 will be used to capture 3 x 24-hour dietary intake recalls at baseline and endpoint to assess changes in dietary protein measured in grams (g). This is a validated web-based 24-hour dietary assessment tool for measuring dietary intake.
Change from Baseline in Dietary Energy on 24-hour Dietary Intake Recall at Week 12. | Baseline and Week 12.
  Intake24 will be used to capture 3 x 24-hour dietary intake recalls at baseline and endpoint to assess changes in dietary energy measured in kilocalories (kcal). This is a validated web-based 24-hour dietary assessment tool for measuring dietary intake.
Apolipoprotein E (APOE) and Fatty Acid Desaturase (FADS) Genotypes. | Baseline.
  ApoE and FADs genotypes will be measured.
Change from Baseline in Dietary Long-Chain Omega-3 Polyunsaturated Fatty Acids (LCn-3 PUFA) Intake at Week 12. | Baseline and Week 12.
  LCn-3 PUFA dietary intake changes will be assessed with a validated food frequency questionnaire (FFQ).
Change from Baseline in Whole Blood Fatty Acid Profile at Week 12. | Baseline and Week 12.
  Whole fatty acid composition will be measured.
Change from Baseline in Glutamate Concentrations in the Right and Left Ventrolateral Prefrontal Cortex and the Anterior Cingulate Cortex at Week 12. | Baseline and Week 12.
  Proton Magnetic resonance spectroscopy will be used to assess neurochemical changes in response to supplementation.
Change from Baseline in Seed-to-Voxel Functional Connectivity using Bilateral Orbitofrontal Cortex and Amygdala Seeds at Week 12. | Baseline and Week 12.
  Functional magnetic resonance imaging will be used to assess changes in functional connectivity in response to supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Gibson, PhD, Study Director — University of Roehampton; Simon Dyall, PhD, Principal Investigator — University of Roehampton
Locations (1):
- University of Roehampton, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be:
  * Fully anonymised
  * Stored for 8 years as per University of Roehampton's Research Ethics Committee guidelines and Code of Practice.
  * Appended to the final published report as supplemental material.
  * Available from the corresponding author upon request.
  * Handled, processed, stored and destroyed as per Data Protection Act (2018).
  * Collected in Microsoft Excel worksheets in one file per type of experiment including original and normalised values; images/graphs will be stored as .tiff or .jpg files.
  * Held encrypted on password-protected, university-owned drives.
  * Accessible only by the investigators.
  * Submitted for publication within one year.
  * Deposited in a public preprint server (e.g. bioRxiv). Additional files with legends explaining how the data has been saved and described will be prepared to allow replicability.
  All anonymised data volumes are expected to be small. Long-term backup/archiving will utilise secure in-house facilities and cloud-based storage.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available upon publication of the study report and will remain available for eight years in accordance with the University of Roehampton's Research Ethics Code of Practice.
Access Criteria: Fully anonymised data will be available from the corresponding author upon request.

REFERENCES:
- [Background] Gravielle MC. Activation-induced regulation of GABAA receptors: Is there a link with the molecular basis of benzodiazepine tolerance? Pharmacol Res. 2016 Jul;109:92-100. doi: 10.1016/j.phrs.2015.12.030. Epub 2015 Dec 28. PMID 26733466
- [Background] Masand PS, Gupta S. Long-term side effects of newer-generation antidepressants: SSRIS, venlafaxine, nefazodone, bupropion, and mirtazapine. Ann Clin Psychiatry. 2002 Sep;14(3):175-82. doi: 10.1023/a:1021141404535. PMID 12585567
- [Background] Firth J, Teasdale SB, Allott K, Siskind D, Marx W, Cotter J, Veronese N, Schuch F, Smith L, Solmi M, Carvalho AF, Vancampfort D, Berk M, Stubbs B, Sarris J. The efficacy and safety of nutrient supplements in the treatment of mental disorders: a meta-review of meta-analyses of randomized controlled trials. World Psychiatry. 2019 Oct;18(3):308-324. doi: 10.1002/wps.20672. PMID 31496103
- [Background] O' Donovan F, Carney S, Kennedy J, Hayes H, Pender N, Boland F, Stanton A. Associations and effects of omega-3 polyunsaturated fatty acids on cognitive function and mood in healthy adults: a protocol for a systematic review of observational and interventional studies. BMJ Open. 2019 Jun 22;9(6):e027167. doi: 10.1136/bmjopen-2018-027167. PMID 31230010
- [Background] LeBlanc, N. J., Brown, M., & Henin, A. (2020). Anxiety Disorders in Emerging Adulthood. In E. Bui, M. E. Charney, & A. W. Baker (Eds.), (pp. 157-173).
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Kroenke K, Wu J, Yu Z, Bair MJ, Kean J, Stump T, Monahan PO. Patient Health Questionnaire Anxiety and Depression Scale: Initial Validation in Three Clinical Trials. Psychosom Med. 2016 Jul-Aug;78(6):716-27. doi: 10.1097/PSY.0000000000000322. PMID 27187854
- [Background] Mathias RA, Pani V, Chilton FH. Genetic Variants in the FADS Gene: Implications for Dietary Recommendations for Fatty Acid Intake. Curr Nutr Rep. 2014 Jun;3(2):139-148. doi: 10.1007/s13668-014-0079-1. PMID 24977108
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kiecolt-Glaser JK, Belury MA, Andridge R, Malarkey WB, Glaser R. Omega-3 supplementation lowers inflammation and anxiety in medical students: a randomized controlled trial. Brain Behav Immun. 2011 Nov;25(8):1725-34. doi: 10.1016/j.bbi.2011.07.229. Epub 2011 Jul 19. PMID 21784145
- [Background] McNamara RK, Strawn JR, Tallman MJ, Welge JA, Patino LR, Blom TJ, DelBello MP. Effects of Fish Oil Monotherapy on Depression and Prefrontal Neurochemistry in Adolescents at High Risk for Bipolar I Disorder: A 12-Week Placebo-Controlled Proton Magnetic Resonance Spectroscopy Trial. J Child Adolesc Psychopharmacol. 2020 Jun;30(5):293-305. doi: 10.1089/cap.2019.0124. Epub 2020 Mar 11. PMID 32167792
- [Background] McNamara RK, Li W, Lei D, Tallman MJ, Welge JA, Strawn JR, Patino LR, DelBello MP. Fish oil supplementation alters emotion-generated corticolimbic functional connectivity in depressed adolescents at high-risk for bipolar I disorder: A 12-week placebo-controlled fMRI trial. Bipolar Disord. 2022 Mar;24(2):161-170. doi: 10.1111/bdi.13110. Epub 2021 Jul 23. PMID 34214231
- [Derived] Kelaiditis CF, Gibson EL, Dyall SC. The effects of a high eicosapentaenoic acid multinutrient supplement on measures of stress, anxiety and depression in young adults: Study protocol for NutriMOOD, a randomised double-blind placebo-controlled trial. Prostaglandins Leukot Essent Fatty Acids. 2021 Oct;173:102335. doi: 10.1016/j.plefa.2021.102335. Epub 2021 Aug 25. PMID 34461561